CLINICAL TRIAL: NCT02654067
Title: Evaluation of Mallampati Score Changes in Pregnancy
Status: Withdrawn | Type: Observational
Why Stopped: Lack of available personnel to conduct data acquisition and analysis
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Julian N Robinson, Chief of Obstetrics, Brigham and Women's Hospital
Other Study IDs: Pregnancy Airway Study
Record Dates: First submitted 2015-11-25; First posted 2016-01-13 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Pregnancy
MeSH Terms: interventions — Moire Topography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: photograph — photograph of airway

SUMMARY:
Pregnant patients mallampati class scores will be examined throughout pregnancy

DETAILED DESCRIPTION:
Photographs of the airway will be taken and compared throughout labor and delivery

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* at least 18 years of age

Exclusion Criteria:

* refusal of consent
* known difficult airway

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mallampati score changes during pregnancy | 40 weeks
  mallampati scores classification from 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Julian Robinson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Mallampati SR, Gatt SP, Gugino LD, Desai SP, Waraksa B, Freiberger D, Liu PL. A clinical sign to predict difficult tracheal intubation: a prospective study. Can Anaesth Soc J. 1985 Jul;32(4):429-34. doi: 10.1007/BF03011357. PMID 4027773
- [Result] Kodali BS, Chandrasekhar S, Bulich LN, Topulos GP, Datta S. Airway changes during labor and delivery. Anesthesiology. 2008 Mar;108(3):357-62. doi: 10.1097/ALN.0b013e31816452d3. PMID 18292672
- [Result] Pilkington S, Carli F, Dakin MJ, Romney M, De Witt KA, Dore CJ, Cormack RS. Increase in Mallampati score during pregnancy. Br J Anaesth. 1995 Jun;74(6):638-42. doi: 10.1093/bja/74.6.638. PMID 7640115